CLINICAL TRIAL: NCT01138553
Title: A Biomarker Study of Mifepristone in Early Stage Breast Cancer
Brief Title: Preoperative Testing of the Anti-Progesterone Mifepristone in Early Stage Breast Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inadequate subject accrual
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard Schwab, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD#100231
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Invasive Breast Cancer; Ductal Carcinoma in Situ
Keywords: biomarker; breast cancer; antiprogesterone
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mifepristone (Experimental)
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — 200mg capsules daily for 5-28 days

SUMMARY:
The primary objective of this study is to identify the group of women with early stage breast cancer most likely to benefit from treatment with the selective progesterone receptor modulator (SPRM) mifepristone. This will be done by treating women briefly prior to planned surgery and examining the decrease in growth rate (measured by Ki-67 immunohistochemistry) in tumor samples taken before and after exposure to mifepristone.

DETAILED DESCRIPTION:
Secondary objectives of this study include; (1) Measuring objective response in tumor size with treatment, (2) Establishing the safety and tolerability of short term mifepristone exposure in early stage breast cancer patients, and (3) Performing exploratory studies of expression of related targets following drug exposure.

Anti-estrogen therapy has been a mainstay of breast cancer treatment for over three decades. It is highly effective and has modest toxicity, certainly in comparison to chemotherapy. The selective estrogen receptor modulator tamoxifen has the longest history but a number of aromatase inhibitors and the anti-estrogen fulvestrant are also in widespread use along with ovarian ablation for pre-menopausal women. Given the success of this approach, and the highly analogous parallel progesterone signal, it is unfortunate that anti-progesterone therapy has not been similarly pursued. Additionally, data from the Woman's Health Initiative trial reveal a potentially significant role for progesterone in breast cancer development and growth. Healthy postmenopausal women treated with the combination of estrogen and progesterone over a 5 year period were 24% more likely to develop invasive breast cancer and had larger tumors at diagnosis. Notably this effect was not seen in post-hysterectomy women treated with estrogen alone over nearly 7 years. In fact a non-statistically significant reduction in breast cancer incidence was observed with estrogen alone.

The anti-progesterone mifepristone has been found to reduce proliferation in normal breast tissue. Even a low dose of mifepristone (50mg every other day for 3 months) demonstrated a statistically significant reduction in breast cell proliferation (measured by Ki-67 immunohistochemistry).

Higher doses of mifepristone, 200mg daily, have been used in patients with metastatic breast cancer for durations of almost 2 years without serious toxicity. Response rates were only 11% but no grade 4 or 5 toxicities occurred. Some grade 3 toxicities occurred, including lethargy, nausea, vomiting, and skin rash. These rashes resolved with temporary discontinuation of drug and did not recur when drug was resumed.

As a whole these data strongly support research into anti-progesterone therapy for early stage breast cancer. To our knowledge this is the first such study.

ELIGIBILITY:
Inclusion Criteria:

* Female identified as a candidate for primary resection of breast cancer (invasive or ductal carcinoma in situ) by a UCSD Breast Care Unit surgical oncologist
* Subjects must agree to contact the study coordinator prior to starting any new medications, vitamins or herbals during, or for 2 weeks following, mifepristone use
* Subjects must agree to abstain from alcohol use while on mifepristone
* Age ≥18
* ECOG performance status 0-1
* Prior to starting mifepristone subjects must have a negative urine (βHCG combo with on-board control) or blood pregnancy test and must be using one of the following acceptable means of birth control prior to starting study drug; Barrier methods or surgically sterile (tubal ligation, hysterectomy or partner with confirmed vasectomy). Alternatively the subject must be one year post-menopausal defined as greater than 12 months without a menstrual cycle
* Prior to starting mifepristone subjects must meet the following laboratory criteria; Granulocytes > 1.5E9/l (grade ≤ 1); Platelets ≥ 100E9/l; Hemoglobin > 10 g/dl (grade ≤ 1); Creatinine < 1.5x normal reference range (grade ≤ 1); SGOT, SGPT, alk phos ≤ 1x normal reference range; Total bilirubin < 1x normal reference range; Calcium < 11.5 mg/dl (grade ≤ 1); HBsAg = Negative; HCV Ab = Negative; INR < 1.5;
* Subjects must provide written informed consent

Exclusion Criteria:

* Not scheduled for surgery within 5 days of enrollment
* Subjects must not be on any therapy to treat breast cancer prior to surgical resection, specifically medications or recent (within 1 month of diagnostic biopsy) withdrawal of estrogen containing medication (eg. hormone replacement therapy)
* Subjects must not be on any medications, vitamins or herbals that are; potent inhibitors of cytochrome P450 CYP3A4, or sensitive substrates for cytochrome P450 CYP3A4
* Subjects may not have any history of significant cardiovascular, renal or hepatic disease requiring ongoing medical therapy or clinical intervention
* Subjects may not have a history of thrombophlebitis, thromboembolic disorder, or cerebral vascular disease.
* Subjects may not have any known hypersensitivity to mifepristone
* Subjects may not have a BMI > 39
* Subjects may not have an IUD (Intrauterine contraceptive device), chronic adrenal failure, concurrent long term steroid therapy, history of allergy to mifepristone, hemorrhagic disorders or concurrent anticoagulant therapy, or inherited porphyrias

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in proliferation by Ki-67 immunohistochemistry. | 5-30 days

SECONDARY OUTCOMES:
Tumor size | 5-30 days
Expression of related targets following mifepristone exposure | 5-28 days
  RNA-seq will be used to evaluate expression of steroid receptor isoform expression following drug exposure. These data will be compared with response as measured by proliferation change and tumor size.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Schwab, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Background] Chlebowski RT, Hendrix SL, Langer RD, Stefanick ML, Gass M, Lane D, Rodabough RJ, Gilligan MA, Cyr MG, Thomson CA, Khandekar J, Petrovitch H, McTiernan A; WHI Investigators. Influence of estrogen plus progestin on breast cancer and mammography in healthy postmenopausal women: the Women's Health Initiative Randomized Trial. JAMA. 2003 Jun 25;289(24):3243-53. doi: 10.1001/jama.289.24.3243. PMID 12824205
- See also: UCSD Moores Cancer Center Clinical Trials — http://cancer.ucsd.edu/clinical-trials/Pages/search.aspx